CLINICAL TRIAL: NCT07312071
Title: Vasopressor Use Improves Macrocirculation, But What Are Its Effects on Microcirculation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Oguz Özakın, Anesthesiology and Reanimation Specialist, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1234
Record Dates: First submitted 2023-07-07; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock; Sepsis; Tissue Ischemia; Hemodynamic Instability
Keywords: Tissue oxygenation; Vazopressor; Septic Shock; Sepsis; microcirculation
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other): The study will include adult patients aged 18 and above who are receiving vasopressor therapy due to septic shock in the intensive care unit.
  Interventions: Diagnostic Test: Vascular Occlusion Test

INTERVENTIONS:
Diagnostic Test: Vascular Occlusion Test — The vascular occlusion test is a procedure performed to assess the vascular status and perfusion of a limb. It involves temporarily stopping blood flow to the limb by applying a blood pressure cuff.

SUMMARY:
To manage the treatment in the intensive care unit for patients with septic shock, central venous oxygen saturation (scvO2) is used as a macrocirculatory indicator, with a target value of 70% or higher being recommended. Tissue oxygenation (stO2) measurement can be implemented to assess the microcirculation in these patients, but a specific target value has not been established yet. The investigators believe that guiding the treatment of septic shock patients based on the measurement of microcirculation using stO2 and evaluating its correlation with scvO2 can reduce mortality.

This study aims to investigate the independent impact of high-dose norepinephrine on microvascular reactivity assessed by NIRS-VOT in patients with septic shock, while also examining how these microcirculatory indices relate to the macrocirculatory marker ScvO₂.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of septic shock
* Receiving vasopressor and mechanical ventilation therapy
* Presence of a central venous catheter that allows ScvO₂ sampling
* Ability to obtain tissue oxygenation (stO₂) measurements using a NIRS probe placed on the thenar eminence
* Written informed consent obtained from patient or legal representative

Exclusion Criteria:

* Local infection, wound, or skin lesion at the planned NIRS probe application site
* Mean arterial pressure (MAP) < 60 mmHg despite vasopressor therapy
* Pregnancy
* Inability to safely perform the vascular occlusion test (as judged by treating clinician)
* Any condition preventing safe blood sampling or reliable stO₂ measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Central Venous Oxygen Saturation (ScvO₂) Level | Baseline (first 1 hour)
  Central venous oxygen saturation will be measured from a central venous blood gas sample. The ScvO₂ value obtained at baseline will be recorded.
Norepinephrine Equivalent Vasopressor Dose | Baseline (first 1 hour)
  The vasopressor requirement will be expressed as the norepinephrine equivalent dose (NEq), calculated in µg/kg/min.
Baseline Tissue Oxygen Saturation (stO₂_baseline) | Within 1 hour of enrollment
  Tissue oxygen saturation will be measured non-invasively from the thenar eminence using Near-Infrared Spectroscopy (NIRS). The baseline stO₂ value will be recorded immediately before the vascular occlusion test.
Minimum Tissue Oxygen Saturation During Vascular Occlusion (stO₂_min) | Within 1 hour of enrollment
  During the vascular occlusion test (inflation of a cuff to stop arterial inflow), the lowest tissue oxygen saturation (stO₂_min) recorded from the NIRS probe on the thenar eminence will be measured and recorded.
Maximum Tissue Oxygen Saturation After Reperfusion (stO₂_max) | Within 1 hour of enrollment
  After release of the vascular occlusion, the highest tissue oxygen saturation (stO₂_max) value recorded during reactive hyperemia will be measured and recorded.
Recovery Time (From stO₂_min to stO₂_max) | Within 1 hour of enrollment
  Recovery time will be defined as the time interval between the minimum tissue oxygen saturation (stO₂_min) during vascular occlusion and the maximum tissue oxygen saturation (stO₂_max) after cuff release, as measured by NIRS on the thenar eminence.

SECONDARY OUTCOMES:
28-Day All-Cause Mortality | 28 days
  Vital status (alive or deceased) will be assessed 28 days after enrollment to determine all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided